CLINICAL TRIAL: NCT00603226
Title: Slow Coronary Artery Flow: Influence on Morbidity and Mortality
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Yaniv Levi, Hillel Yaffe Medical Center
Other Study IDs: 57/2007
Record Dates: First submitted 2008-01-16; First posted 2008-01-29 (Estimated); Last update posted 2008-01-29 (Estimated); Status verified 2008-01

CONDITIONS: Coronary Disease
Keywords: Coronary slow flow phenomenon; Coronary angiography; Acute coronary syndrome; Chest pain; Unstable angina
MeSH Terms: conditions — Coronary Disease; Acute Coronary Syndrome; Chest Pain; Angina, Unstable

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Patients diagnosed with slow coronary artery flow during coronary angiography
- 2: Patients with normal coronary artery flow observed during coronary angiography

SUMMARY:
To compare patients with Slow Coronary Artery Flow to patients with normal flow and to determine whether there is a difference in their future incidence of heart disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent coronary angiography

Exclusion Criteria:

* Patients with coronary occulsion above 50%
* Patients with severe valve disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent coronary angiography in the Hillel Yaffe Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2008-01; Primary Completion 2008-07 (Estimated); Study Completion 2008-07 (Estimated)

PRIMARY OUTCOMES:
How many hospitalizations for major coronary events in patients with or without slow coronary artery flow. | Six months

CONTACTS AND LOCATIONS:
Overall Officials: Yaniv Levi, MD, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel